## The SAFE Study: <u>Satisfaction and Adherence to Follow-Up with</u> Colposcopy <u>Exams</u>

**Statistical Analysis Plan** 

SAFE #H16-03194 NCT03296566 v.1 2020-03-30 We compared demographic and clinical baseline variables between the groups using Wilcoxon rank-sum tests for continuous variables and Fisher's exact tests for categorical variables. We compared age, education, employment, and pathology results between those who completed the survey and those who did not using Wilcoxon rank-sum tests for continuous variables and Fisher's exact tests for categorical variables.

The primary outcome (STAI - STATE scores) was compared between the groups using a t-test. Secondary outcomes were compared between the groups using t-tests for continuous variables and Fisher's exact tests for categorical variables. We also built a multiple linear regression model to examine the difference between the groups in STAI-STATE scores while controlling for STAI-TRAIT scores and the severity of the diagnosis (Negative, CIN 1, CIN 2, and CIN 3). One case of serous carcinoma was included in the CIN 3 category.